CLINICAL TRIAL: NCT05631119
Title: Biorepository of Biospecimen Samples in Matched Healthy Control Participants and Participants Diagnosed With Diabetic Kidney Disease, Chronic Kidney Disease, or Type 2 Diabetes
Acronym: SAN-08961
Status: Completed | Type: Observational
Sponsor: Sanguine Biosciences (Industry)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: SAN-08961
Record Dates: First submitted 2022-11-15; First posted 2022-11-30 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Diabetic Kidney Disease; Diabetes Type 2; Chronic Kidney Diseases; Healthy
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Diabetic Kidney Disease: Sample Collection:
  * Whole blood will be collected in 3 x 5 mL SST tubes. The samples will be centrifuged into 5 x 1 mL serum aliquots. The aliquots will be shipped frozen (with dry ice) overnight to Novo Nordisk via FedEx Priority Overnight by 10:30 am.
  * Whole blood will be collected in 4 x 10 mL and 1 x 4 mL sodium heparin tubes. The samples will be shipped ambient overnight to Sanguine Labs via FedEx Priority Overnight by 10:30 am. Sanguine Labs will process the samples for PBMC isolations at 10 million cells per aliquot. Samples will be stored for batch shipment at the end of the study. The PBMC aliquot(s) will be shipped overnight using liquid nitrogen (LN2) to Novo Nordisk via FedEx Priority Overnight by 10:30 am.
  * Urine will be collected using a Vacuette collection device. The sample will be shipped frozen (with dry ice) overnight to Novo Nordisk via FedEx Priority Overnight by 10:30
- Chronic Kidney Disease: Sample Collection:
  * Whole blood will be collected in 3 x 5 mL SST tubes. The samples will be centrifuged into 5 x 1 mL serum aliquots. The aliquots will be shipped frozen (with dry ice) overnight to Novo Nordisk via FedEx Priority Overnight by 10:30 am.
  * Whole blood will be collected in 4 x 10 mL and 1 x 4 mL sodium heparin tubes. The samples will be shipped ambient overnight to Sanguine Labs via FedEx Priority Overnight by 10:30 am. Sanguine Labs will process the samples for PBMC isolations at 10 million cells per aliquot. Samples will be stored for batch shipment at the end of the study. The PBMC aliquot(s) will be shipped overnight using liquid nitrogen (LN2) to Novo Nordisk via FedEx Priority Overnight by 10:30 am.
  * Urine will be collected using a Vacuette collection device. The sample will be shipped frozen (with dry ice) overnight to Novo Nordisk via FedEx Priority Overnight by 10:30 am
- Type 2 Diabetes: Sample Collection:
  * Whole blood will be collected in 3 x 5 mL SST tubes. The samples will be centrifuged into 5 x 1 mL serum aliquots. The aliquots will be shipped frozen (with dry ice) overnight to Novo Nordisk via FedEx Priority Overnight by 10:30 am.
  * Whole blood will be collected in 8 x 10 mL and 1 x 4 mL sodium heparin tubes. The samples will be shipped ambient overnight to Sanguine Labs via FedEx Priority Overnight by 10:30 am. Sanguine Labs will process the samples for PBMC isolations at 10 mL cells per aliquot. Samples will be stored for batch shipment at the end of the study. The PBMC aliquot(s) will be shipped overnight using liquid nitrogen (LN2) to Novo Nordisk via FedEx Priority Overnight by 10:30 am.
  * Urine will be collected using a Vacuette collection device. The sample will be shipped frozen (with dry ice) overnight to Novo Nordisk via FedEx Priority Overnight by 10:30 am.
- Healthy Matched Controls: Sample Collection:
  * Whole blood will be collected in 3 x 5 mL SST tubes. The samples will be centrifuged into 5 x 1 mL serum aliquots. The aliquots will be shipped frozen (with dry ice) overnight to Novo Nordisk via FedEx Priority Overnight by 10:30 am.
  * Whole blood will be collected in 16 x 10 mL and 1 x 4 mL sodium heparin tubes. The samples will be shipped ambient overnight to Sanguine Labs via FedEx Priority Overnight by 10:30 am. Sanguine Labs will process the samples for PBMC isolations at 10 mL cells per aliquot. Samples will be stored for batch shipment at the end of the study. The PBMC aliquot(s) will be shipped overnight using liquid nitrogen (LN2) to Novo Nordisk via FedEx Priority Overnight by 10:30 am.
  * Urine will be collected using a Vacuette collection device. The sample will be shipped frozen (with dry ice) overnight to Novo Nordisk via FedEx Priority Overnight by 10:30 am.

SUMMARY:
The Investigators will generate a repository of human biosamples across therapeutic areas that will be used to identify disease-associated biomarkers and potential targets with immune and multi-omics profiling. This sample collection and analysis from people living with type 2 diabetes, or chronic or diabetic kidney disease will lay the groundwork for an extensive network of biosample access and linked datasets that will provide an invaluable resource for translational research.

DETAILED DESCRIPTION:
The Investigators will generate a repository of human biosamples across therapeutic areas that will be used to identify disease-associated biomarkers and potential targets with immune and multi-omics profiling. This sample collection and analysis from people living with type 2 diabetes, or chronic or diabetic kidney disease will lay the groundwork for an extensive network of biosample access and linked datasets that will provide an invaluable resource for translational research.

ELIGIBILITY:
Cohort 1: Diabetic Kidney Disease

Inclusion:

1. The participant is willing and able to provide written informed consent
2. The participant is willing and able to provide appropriate photo identification
3. Participants aged 18 to 85
4. Participants have been diagnosed with diabetic kidney disease. Enrollment preference for participants with stage 3 kidney disease but is not inclusionary.

Exclusion:

1. Participants who are pregnant or are nursing
2. Participants with a known history of HIV, hepatitis, or other infectious diseases
3. Participants who have taken an investigational product in the last 30 days
4. Participants who have experienced excess blood loss, including blood donation, defined as 250 mL in the last month or 500 mL in the previous two months

Cohort 2: Chronic Kidney Disease

Inclusion:

1. The participant is willing and able to provide written informed consent
2. The participant is willing and able to provide appropriate photo identification
3. Participants aged 18 to 85
4. Participants have been diagnosed with chronic kidney disease.

Exclusion:

1. Participants who are pregnant or are nursing
2. Participants with a known history of HIV, hepatitis, or other infectious diseases
3. Participants who have taken an investigational product in the last 30 days
4. Participants who have experienced excess blood loss, including blood donation, defined as 250 mL in the last month or 500 mL in the previous two months
5. Participants have been diagnosed with acute kidney disease or diabetic kidney disease

Cohort 3: Type 2 Diabetes

Inclusion:

1. The participant is willing and able to provide written informed consent
2. The participant is willing and able to provide appropriate photo identification
3. Participants aged 18 to 85
4. Participants have been diagnosed with type 2 diabetes.

Exclusion:

1. Participants who are pregnant or are nursing
2. Participants with a known history of HIV, hepatitis, or other infectious diseases
3. Participants who have taken an investigational product in the last 30 days
4. Participants who have experienced excess blood loss, including blood donation, defined as 250 mL in the last month or 500 mL in the previous two months
5. Participants have been diagnosed with type 1 diabetes

Cohort 4: Healthy Matched The study will enroll participants considered healthy matched controls per the eligibility criteria. The healthy-matched controls must match each participant in the diseased cohorts by age (+/- 10 years).

Inclusion:

1. The participant is willing and able to provide written informed consent 2. The participant is willing and able to provide appropriate photo identification 3. Participants aged 18 to 85 4. Participants who are in generally good health are defined as: b. Participants may have a common/mild health condition(s) that are generally under control, including but not limited to: i. Hypertension, high cholesterol, asthma, anxiety, depression, attention deficit disorder (ADD), attention deficit hyperactivity disorder (ADHD), gastroesophageal reflux disease (GERD), irritable bowel syndrome (IBS), allergies, eczema, migraines, osteoarthritis, sleep apnea, restless leg syndrome, and eye issues (e.g., myopia, astigmatism, etc.) ii. Participants with a previous diagnosis and have recovered from COVID-19 iii. Participants in general good health may also take nonsteroidal anti-inflammatory drugs (NSAIDS) (i.e., ibuprofen, Tylenol, aspirin, Excedrin) irregularly or semi-regularly due to conditions like headache, body aches, cold/flu treatment as long as the medications are not being used for the treatment of a major underlying condition.

Exclusion:

1. Participants who are pregnant or are nursing
2. Participants with a known history of HIV, hepatitis, or other infectious diseases
3. Participants who have taken an investigational product in the last 30 days
4. Participants who have experienced excess blood loss, including blood donation, defined as 250 mL in the last month or 500 mL in the previous two months
5. Participants not considered in general good health

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Diabetic Kidney Disease, Chronic Kidney Disease, and Diabetes Type 2. The 4th cohort will be a healthy match cohort of patients: 2 of the disease cohorts will have 3 healthy matched patieints and the final disease cohort (unspecified) will have 4 healthy patients matched.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-08-23 (Actual); Study Completion 2023-08-23 (Actual)

PRIMARY OUTCOMES:
collect biospecimen samples | 7 months
  The study objective is to collect biospecimen samples (e.g., blood and urine) from participants diagnosed with diabetic kidney disease, chronic kidney disease, or type 2 diabetes. These samples will be used to generate a repository of human biosamples across therapeutic areas that will be used to identify disease-associated biomarkers and potential targets with immune and multi-omics profiling. This sample collection and analysis from people living with type 2 diabetes, or chronic or diabetic kidney disease will lay the groundwork for an extensive network of biosample access and linked datasets that will provide an invaluable resource for translational research.

CONTACTS AND LOCATIONS:
Locations (1):
- Sanguine Biosciences, Inc., Woburn, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] National Institute of Health (NIH): National Center for Advancing Translational Sciences. Understanding Translational Research Tools: Biorepository. Accessed: 19 October 2022. https://toolkit.ncats.nih.gov/module/discovery/developing-translational-research-tools/biorepository/
- [Background] Siwek M. An Overview of Biorepositories-Past, Present, and Future. Mil Med. 2015 Oct;180(10 Suppl):57-66. doi: 10.7205/MILMED-D-15-00119. PMID 26444893
- [Background] Strimbu K, Tavel JA. What are biomarkers? Curr Opin HIV AIDS. 2010 Nov;5(6):463-6. doi: 10.1097/COH.0b013e32833ed177. PMID 20978388
- [Background] Quezada H, Guzman-Ortiz AL, Diaz-Sanchez H, Valle-Rios R, Aguirre-Hernandez J. Omics-based biomarkers: current status and potential use in the clinic. Bol Med Hosp Infant Mex. 2017 May-Jun;74(3):219-226. doi: 10.1016/j.bmhimx.2017.03.003. Epub 2017 May 10. PMID 29382490
- [Background] Kreeger K. Immune Profiling: A New Opportunity for Drug Development. Penn Medicine News. February 14, 2019. Accessed: 20 October 2022. https://www.pennmedicine.org/news/news-blog/2019/february/immune-profiling-a-new-opportunity-for-drug-development
- [Background] Chuah S, Chew V. High-dimensional immune-profiling in cancer: implications for immunotherapy. J Immunother Cancer. 2020 Feb;8(1):e000363. doi: 10.1136/jitc-2019-000363. PMID 32034066
- [Background] Olivier M, Asmis R, Hawkins GA, Howard TD, Cox LA. The Need for Multi-Omics Biomarker Signatures in Precision Medicine. Int J Mol Sci. 2019 Sep 26;20(19):4781. doi: 10.3390/ijms20194781. PMID 31561483
- [Background] Krassowski M, Das V, Sahu SK, Misra BB. State of the Field in Multi-Omics Research: From Computational Needs to Data Mining and Sharing. Front Genet. 2020 Dec 10;11:610798. doi: 10.3389/fgene.2020.610798. eCollection 2020. PMID 33362867
- [Background] Subramanian I, Verma S, Kumar S, Jere A, Anamika K. Multi-omics Data Integration, Interpretation, and Its Application. Bioinform Biol Insights. 2020 Jan 31;14:1177932219899051. doi: 10.1177/1177932219899051. eCollection 2020. PMID 32076369
- [Background] Khan MAB, Hashim MJ, King JK, Govender RD, Mustafa H, Al Kaabi J. Epidemiology of Type 2 Diabetes - Global Burden of Disease and Forecasted Trends. J Epidemiol Glob Health. 2020 Mar;10(1):107-111. doi: 10.2991/jegh.k.191028.001. PMID 32175717
- [Background] Roy S, Schweiker-Kahn O, Jafry B, Masel-Miller R, Raju RS, O'Neill LMO, Correia CR, Trivedi A, Johnson C, Pilot C, Saddemi J, Memon A, Chen A, McHugh SP, Patel S, Daroshefski NM, Nguyen T, Wissler W, Sharma E, Hunter K. Risk Factors and Comorbidities Associated with Diabetic Kidney Disease. J Prim Care Community Health. 2021 Jan-Dec;12:21501327211048556. doi: 10.1177/21501327211048556. PMID 34634970
- [Background] Garcia-Carro C, Vergara A, Bermejo S, Azancot MA, Sanchez-Fructuoso AI, Sanchez de la Nieta MD, Agraz I, Soler MJ. How to Assess Diabetic Kidney Disease Progression? From Albuminuria to GFR. J Clin Med. 2021 Jun 5;10(11):2505. doi: 10.3390/jcm10112505. PMID 34198818